CLINICAL TRIAL: NCT05574257
Title: Comparison of the Effect of Remimazolam and Propofol on Perioperative Hypothermia Under Spinal Anesthesia: A Randomized Control Study.
Brief Title: Comparison of the Effect of Remimazolam and Propofol on Perioperative Hypothermia Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor of Anesthesiology and Pain Medicine, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WonkwangUH12
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Lower Extremity Problem; Gynecologic Disease; Urinary Tract Disease
MeSH Terms: conditions — Genital Diseases, Female; Urologic Diseases | interventions — Propofol; remimazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): The group received propofol injection at 25-100ug/kg/min (immediately after spinal anesthesia to the end of surgery).
  Interventions: Drug: Propofol
- Group R (Experimental): The group received remimazolam injection at 1-20ug/kg/min (immediately after spinal anesthesia to the end of surgery).
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Propofol — Propofol is injected at 25-100ug/kg/min (immediately after spinal anesthesia to the end of surgery) to maintain the BIS at 70-80.
  Other Names: Fresofol®
  Arms: Group P
Drug: Remimazolam — Remimazolam is injected at 1-20ug/kg/min (immediately after spinal anesthesia to the end of surgery) to maintain the BIS at 70-80.
  Other Names: Byfavo®
  Arms: Group R

SUMMARY:
After dividing the patients into two groups, sedation is performed with propofol and remimazolam, respectively, after spinal anesthesia. Compare the patient's body temperature change after surgery.

DETAILED DESCRIPTION:
Patients in the study were randomly assigned to the propofol group (Group P) and the remimazolam group (Group R) in a 1:1 ratio. Study drugs are prepared in the same 50 ml syringe, double-blind to group assignment. All patients are not given pre-anesthetic medication, and body temperature, blood pressure, and heart rate are measured in the recovery room after surgery at 10-minute intervals from just before anesthesia induction to surgery. If hypotension or bradycardia occurs during surgery and is not corrected even after rapid fluid infusion, ephedrine is increased by 10 mg or glycopyrrolate 0.2 mg or atropine 0.5 mg is administered.

If spinal anesthesia is successfully performed, check the patient's anesthesia height. When the appropriate level of anesthesia is confirmed, Group P receives propofol at 25-100ug/kg/min and maintains the BIS at 70-80. Group R receives remimazolam at 1-20ug/kg/min and maintains BIS between 70-80. Both groups apply a conventionally used air heating device, and the operating room temperature is kept at 20 °C. If shivering occurs during surgery, the elapsed time from induction and the shivering grades are recorded.

At the end of the surgery, record total anesthesia time and surgery time, fluid dose, and drug use. After moving to the recovery room, the patient's body temperature, systolic blood pressure, diastolic pressure, heart rate, the incidence of shivering, and the grade of shivering are checked. When shivering occurs, a forced air-warming device is applied first, and if shivering continues, administer meperidine in 5mg increments until the patient is comfortable and record the total dose.

ELIGIBILITY:
Inclusion Criteria:

* Those aged between 19 and under 65 who are undergoing surgery under spinal anesthesia at Wonkwang University Hospital.
* American Society of Anesthesiologists' physical status class (ASA) award class I-III.

Exclusion Criteria:

* Patients with fever before surgery
* Patients taking antipyretics before surgery
* Patients who are chronically using anti-inflammatory drugs
* High-risk patients with ASA class IV or higher
* Patient who refused sedation
* Patients with thyroid dysfunction.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
The incidence of perioperartive hypothermia | During surgery
  Measure the body temperature on the tympanic membrane three times and enter the highest value.
The incidence of perioperartive hypothermia | At PACU (Post Anesthesia Care Unit)
  measure the body temperature three times on the tympanic membrane and enter the highest value.

SECONDARY OUTCOMES:
core body temperature | Before the induction of anesthesia
  Every 10 minutes, measure the body temperature three times on the tympanic membrane and enter the highest value.
core body temperature | During surgery
  Every 10 minutes, measure the body temperature three times on the tympanic membrane and enter the highest value.
core body temperature | At PACU
  Every 10 minutes, measure the body temperature three times on the tympanic membrane and enter the highest value.
shivering grades | During surgery
  1. None (Grade 0): no shivering noted on palpation of the masseter, neck, or chest wall
  2. Mild (Grade 1): shivering localized to the neck and/or thorax only
  3. Moderate (Grade 2): shivering involved the gross movement of the upper extremities (in addition to neck and thorax)
  4. Severe (Grade 3): shivering involved gross trunk and upper and lower extremities movements.
shivering grades | At PACU
  1. None (Grade 0): no shivering noted on palpation of the masseter, neck, or chest wall
  2. Mild (Grade 1): shivering localized to the neck and/or thorax only
  3. Moderate (Grade 2): shivering involved the gross movement of the upper extremities (in addition to neck and thorax)
  4. Severe (Grade 3): shivering involved gross trunk and upper and lower extremities movements.

CONTACTS AND LOCATIONS:
Overall Officials: Cheolhyeong Lee, M.D., Principal Investigator — Wonkwang University Hospital
Locations (1):
- Wonkwag UH, Iksan, Jeollabukdo, South Korea

IPD SHARING:
Plan to Share IPD: No